CLINICAL TRIAL: NCT01411124
Title: A Randomized, Double-Blind, Active- and Placebo-Controlled, Crossover Study Assessing the Effect of 600 mg Gabapentin Enacarbil on Simulated Driving in Healthy Subjects
Brief Title: Study to Assess the Effect of Gabapentin Enacarbil on Simulated Driving in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114111
Record Dates: First submitted 2011-07-28; First posted 2011-08-08 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2011-11

CONDITIONS: Restless Legs Syndrome (RLS)
Keywords: gabapentin; restless leg syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gabapentin Enacarbil (Experimental): 600 mg of Gabapentin Enacarbil
  Interventions: Drug: gabapentin enacarbil; Drug: placebo
- diphenhydramine (Active Comparator): 50 mg
  Interventions: Drug: diphenhydramine; Drug: placebo
- placebo (Placebo Comparator): placebo to match
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: gabapentin enacarbil — 600 mg investigational compound
  Other Names: XP13512; GSK1838262
  Arms: Gabapentin Enacarbil
Drug: diphenhydramine — 50 mg active comparator
  Arms: diphenhydramine
Drug: placebo — placebo

SUMMARY:
This is a double-blind, placebo-and active-controlled 3-period crossover study designed to assess the effect of GEn 600 mg on simulated driving performance in healthy volunteers.

DETAILED DESCRIPTION:
proportional systemic gabapentin exposure over a wide dose range. This is a double-blind, placebo-and active-controlled 3-period crossover study designed to assess the effect of GEn 600 mg on simulated driving performance. Subjects will receive each of 3 treatments in a randomized order: GEn 600 mg, placebo and placebo/diphenhydramine 50 mg. Each treatment period will consist of 6 days, with subjects being dosed at approximately 5 pm on each dosing day. The placebo /diphenhydramine treatment will consist of placebo on Days 1-4 and 6 and 50 mg diphenhydramine on Day 5. Placebo will be administered on Day 6 in all treatment periods to ensure washout of drug prior to the start of the next treatment period. Simulated driving performance will be assessed at baseline (prior to randomization) and on Day 5 in the evening (7-9 pm) and on Day 6 between7-9 am and between 11am-1pm for each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male or female between 18 and 65 years of age, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation at least 6 months previously or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit is completed.
* Body weight > 50 kg and Body Mass Index (BMI) within the range 19 - 30 kg/m2 (inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* QTcB < 450 msec
* Creatinine clearance (CrCl) >80 mL/min. CrCl is estimated using the equation of Cockcroft and Gault. See study procedure manual for details on creatinine clearance calculations.
* AST, ALT, alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Currently a licensed, experienced driver who drives at least 3 times a week for the past 3 years and with visual acuity assessed by the investigator as being adequate for driving
* Able to complete a 1 hour simulated driving test and demonstrate satisfactory driving skills at screening

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* History of sensitivity to gabapentin, DPH or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive serum human chorionic gonadotrophin (hCG) test at screening or prior to dosing
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* The subject has a screening heart rate <50 or >100 bpm or a systolic blood pressure >140 or <100 mmHg or a diastolic blood pressure >90 or <60 mmHg in the semi-supine position after at least 3 minutes of rest.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease
* History of seizures other than febrile seizures as a child
* Subjects who have received any medications known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration, in the opinion of the Sponsor or Investigator
* Subjects with a creatine kinase (CK) value of greater than the upper limit of normal that is not explainable by recent strenuous exercise and the value does not return within normal range upon retest
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subject is mentally or legally incapacitated
* Subjects with a sleep disorder e.g. sleep apnea, narcolepsy or primary insomnia
* Shift workers who are not on normal day/night sleep cycles
* Subjects with a history of closed angle glaucoma, urinary retention or other conditions for which DPH is contra-indicated
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt
* Subjects who have consumed an average of > 5 cups of caffeinated beverages per day within 20 days of the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Lane performance Variability | From Day-1 baseline to end of treatment. Participants will be followed for the duration of the clinic visit an average of 3 weeks.
  change from baseline in lane position variability

SECONDARY OUTCOMES:
Change in Speed Variability | from baseline to end of treatment Participants will be followed for the duration of the clinic visit an average of 3 weeks
  Change from baseline in speed variability
number of simulated crashes | on Days 5 and 6. The subjects will be followed for the duration of the clinic visit an average of 3 week
  number of simulated crashes
Visual Analog Scale | Baseline to end of treatment. The subjects will be followed for the duration of the clinic visit an average of 3 weeks
  Pre driving alterness measured by the Visual analog scale
Visual analog scale on post driving alertness | baseline to days 5 and 6. The subjects will be followed for the duration of the clinic visit an average of 3 weeks
  Post driving alterness measured by visual alterness scale
Visual Analog scale of the difference between pre and post driving alertness | baseline to days 5 and 6. The subjects will be followed for the duration of the clinic visit an average of 3 weeks
  difference between pre and post driving alertness
Incidents of Adverse events | baseline to end of study. The subjects will be followed for the duration of the clinic visit an average of 3 weeks
  safety and tolerability from baseline to end of study
Plasma concentrations of gabapentin | Day 5. The subjects will be followed for the duration of the clinic visit an average of 3 weeks
  Plasma concentration of gabapentin on completion of driving test

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States